CLINICAL TRIAL: NCT03748927
Title: A Natural History Study of Children and Adults With Fibrolamellar Hepatocellular Carcinoma
Brief Title: Natural History Study of Children and Adults With Fibrolamellar Hepatocellular Carcinoma
Status: Withdrawn | Type: Observational
Why Stopped: slow/insufficient accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190021; 19-C-0021
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer
Keywords: Clinical Outcome; Advice in the Management of Cancer; Patterns of Disease Progression; Response or Lack of Response to Therapeutic Interventions
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1/ Cohort 1: Subjects with FL-HCC.

SUMMARY:
Background:

Fibrolamellar Hepatocellular Carcinoma (FL-HCC) is a rare liver cancer. It usually occurs in young people who have no history of liver disease. Currently the only effective treatment option is surgery that removes the tumor and part of the liver. Researchers want to study the course of the disease to learn more about it.

Objective:

To collect samples from people with FL-HCC to learn more about the disease and help develop new treatments.

Eligibility:

People any age with FL-HCC

Design:

Participants must be enrolled on another NIH protocol.

Participants will have at least 1 study visit. They will have:

* A medical and cancer history
* A physical exam
* A review of their symptoms and their ability to do normal activities
* Tests to produce images of the body. They may have a scan (CT) that uses a small amount of radiation. Or they may have a scan (MRI) that uses a magnetic field. These will examine the chest, abdomen, and pelvis.
* Blood tests

Researchers will study previous tumor samples if they are available.

If participants come to NIH for visits on other studies, data will be collected about their disease, tests, treatments, and responses. Tumor tissue will be collected if participants are having it taken for a procedure.

All other participants will be contacted to collect this data. They will be contacted once a month for 1 year and 2 times a year after that.

Participants will be asked to contact researchers when their health changes. They may come in for more tests.

DETAILED DESCRIPTION:
Background:

* Fibrolamellar hepatocellular carcinoma (FL-HCC) is a rare hepatocellular carcinoma accounting for 0.5-9% of primary liver cancer in various case series, which is usually not associated with elevated serum alpha fetoprotein (AFP) levels, is enriched in younger age groups, and is not associated with underlying liver disease.
* Reports on the characteristics of patients with FL-HCC as well as predictors of recurrence and survival are scarce, largely due to the rarity of this tumor. The only potentially curative treatment option for FL-HCC patients who have resectable disease is surgery: either liver resection (LR) or liver transplantation (LT). However, disease recurrence after complete surgical resection is high, ranging from 33-100%. The clinical outcome of patients with unresectable disease is suboptimal with median survival of less than 12 months and no patient surviving beyond 5 years.
* The role of neoadjuvant and adjuvant therapies, including systemic chemotherapy, remains poorly defined and has been reported to have only a modest or no therapeutic effect. Platinum-based chemotherapy in pediatric patients with FL-HCC resulted a partial response in 31% of patients on imaging but a 3-year survival of only 22%. To date no targeted therapy has been shown to be of any value in this disease.
* The natural history of FL-HCC varies greatly with most patients surviving only months while others can live with the disease for years. While one cannot exclude an immune or other host component as responsible for the diverse clinical courses, it is also possible that there may be a genetic basis for this phenomenon. A novel somatic recurrent 400 kb deletion on the short arm of chromosome 19, giving rise to an in-frame DNAJB1 PRKACA gene fusion was found in FL-HCC. mTOR signaling is significantly activated in FL-HCC compared to other liver malignancies. A bio-specimen repository will be a major step towards more comprehensive studies of this very rare and unusual tumor and allow us to begin to characterize subgroups within the disease.
* Patients with rare tumors seek expert advice in the management of their care. A natural history study would establish a more formal mechanism for such referrals, while allowing the systematic collection of epidemiologic data as well as much needed tumor samples.

Objective:

- Characterize the natural history of Fibrolamellar hepatocellular carcinoma (FL-HCC), including clinical presentation, family history, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival.

Eligibility:

- Subjects of all ages with histologically or cytologically proven FL-HCC.

Design:

* Participants will undergo a comprehensive study entry evaluation including clinical phenotyping and imaging of tumor sites. Computed tomography scans of the thorax, abdomen and pelvis may be performed if clinically indicated; occasionally, magnetic resonance imaging may be performed for the visualization of lesions in the liver, spine, or other anatomic sites if clinically indicated.
* Medical histories will be documented, and participants will be followed throughout the course of their illnesses, with attention to patterns of disease recurrence and progression, response to therapies and duration of responses. As part of this natural history study, growth rates of target tumor lesions will also be calculated throughout the course of the disease whenever available.
* Blood and tumor samples will be obtained at study entry and while on study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects enrolled on NCI protocol Natural History and Biospecimen Acquisition Study for Children and Adults with Rare Solid Tumors
* Subjects of all ages with histologically or cytologically proven FL-HCC.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

None

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Characterize the natural history of Fibrolamellar hepatocellular carcinoma (FL- HCC), including clinical presentation, family history, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurre... | 10 years
  Characterize the natural history of Fibrolamellar hepatocellular carcinoma (FL- HCC), including clinical presentation, family history, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0021.html